CLINICAL TRIAL: NCT05820464
Title: Diastolic Deceleration Area in Severe Early-onset Growth Restriction of the Fetus
Brief Title: Diastolic Deceleration Area in Early-onset FGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Orthogyn Medical Center, Bulgaria (Other)
Responsible Party: Principal Investigator, Petar Ignatov, Assoc. prof. Petar Ignatov, M.D., Ph. D., Orthogyn Medical Center, Bulgaria
Other Study IDs: DDA1
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hypoxia; Anemia
MeSH Terms: conditions — Hypoxia; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Standard care:
  * Doppler velocimetry: UA & MCA PI, DV PIV, CPR;
  * Indirect cardiotocography (CTG)
  * Biophysical profile (BPP)
- DDA Doppler group: Standard care plus DDA Doppler monitoring
  Interventions: Diagnostic Test: DDA Doppler

INTERVENTIONS:
Diagnostic Test: DDA Doppler — A new Doppler parameter to quantify the amount of vasodilatation in the middle cerebral artery (MCA) and other blood vessels.
  Groups: DDA Doppler group

SUMMARY:
DDA is a new Doppler parameter aiming to assess fetal well-being in-utero. Early-onset SGR is a specific subgroup of fetuses where the clinical application of this Doppler modality could play an important role in the detection of hypoxia, anemia, and brain-sparing.

ELIGIBILITY:
Inclusion Criteria:

* absence of fetal abnormalities and/or genetic conditions;
* single pregnancy;
* fetal growth restriction (FGR) < 10%, according to the INTERGROWTH 21st nomograms, appearing before 32nd week of gestation

Exclusion Criteria:

* documented fetal abnormalities and/or genetic conditions in the course of the pregnancy;
* multiple pregnancy;
* absence of fetal growth restriction (FGR) < 10%, according to the INTERGROWTH 21st nomograms before 32nd week of gestation

Ages: 18 Years to 48 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant subjects only
Study Population: No specific criteria, apart from the listed inclusion/exclusion ones
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Hypoxia in the newborn | immediately after delivery
  Defined by pH values below 7.20 in the umbilical artery
Anemia in the newborn | immediately after delivery
  Hemoglobin deviation from GA mean - mild < 20 g/L, moderate - 20-70 g/L, severe > 70 g/L
Occurence of hypoxic-ischemic encephalopathy | first 72 hours after delivery
  Occurence of hypoxic-ischemic encephalopathy in relation to some of the outcome measures

SECONDARY OUTCOMES:
Apgar score at 1st minute | 1 minute after delivery
  Apgar score measured at 1st minute after delivery. Scores ranging from 1 to 10, with higher scores meaning a better outcome.
Apgar score at 5th minute | 5 minutes after delivery
  Apgar score measured at 5th minute after delivery. Scores ranging from 1 to 10, with higher scores meaning a better outcome.
Apgar score at 10th minute | 10 minutes after delivery
  Apgar score measured at 10th minute after delivery. Scores ranging from 1 to 10, with higher scores meaning a better outcome.
Admissions to a NICU | first 72 hours after delivery
  Admissions to a NICU indicated by or related to some of the outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Petar N Ignatov, PhD, Principal Investigator — Orthogyn Medical Center
Locations (1):
- Orthogyn Medical and Dental Center, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided